CLINICAL TRIAL: NCT01304771
Title: A Phase I Trial of the Safety and Efficacy of Adjuvant AKSB (Agri-King Synbiotic) Synbiotic in Patients 65 Years of Age and Older Receiving the Influenza Vaccine
Brief Title: Safety of Synbiotics as Adjuvant to Influenza Vaccine in Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Abinash Virk, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 10-001923; R21AT002708-01A1 (NIH)
Record Dates: First submitted 2010-12-03; First posted 2011-02-25 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Influenza
Keywords: Safety; AKSB; probiotic; synbiotic; enterococcus; Saccharomyces; elderly; influenza; vaccine; immune; response
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Synbiotic AKSB (Active Comparator): Participants (healthy > 65 year old persons) will be randomized to take the synbiotic AKSB. All participants will also receive inactivated trivalent Influenza vaccine while being on the AKSB. We will assess safety of the AKSB in this setting. We will also assess the stool microbiology in relation to vancomycin-resistant enterococcus and probiotic strain enterococcus. We will also assess influenza vaccine response in patients on AKSB
  Interventions: Biological: Synbiotic AKSB
- Talc Placebo (Placebo Comparator): Participants (healthy > 65 year old persons) will be randomized to take the placebo. All participants will also receive inactivated trivalent Influenza vaccine while being on the placebo. We will also assess the stool microbiology in relation to vancomycin-resistant enterococcus. We will also assess influenza vaccine response in patients on placebo.
  Interventions: Biological: Synbiotic AKSB

INTERVENTIONS:
Biological: Synbiotic AKSB — AKSB is a novel synbiotic that contains a probiotic bacterium (Enterococcus faecium, microencapsulated SF68 or Ventrux ME 30), a probiotic yeast (Saccharomyces cerevisiae, Lynside® Pro-Lay 1), and a prebiotic (fructo-oligosaccharide [FOS], NutraFlora®).

SUMMARY:
Probiotics are viable commensal microorganisms that promote the establishment of beneficial microflora. Animal and human studies demonstrate that probiotics can enhance body's immune response to stimuli. Mayo Clinic in conjunction with Agri-King Corporation has developed a novel synbiotic called AKSB (Agri-King Synbiotic) that contains a probiotic bacterium (Enterococcus faecium, microencapsulated SF68 or Ventrux ME 30), a probiotic yeast (Saccharomyces cerevisiae, Lynside® Pro-Lay 1), and a prebiotic (fructo-oligosaccharide [FOS], NutraFlora®). This phase I placebo-controlled trial of AKSB in normal human volunteers, over 65 years of age, is designed to study the safety of this probiotic when patients are also receiving an influenza vaccine. If this study shows that AKSB is safe then our aim is to do a larger study to see if we can improve influenza vaccine immune response while taking the probiotic compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Persons, male and female, 65 years of age and older.
* Eligible and willing to receive the influenza vaccine and take the study drug.
* Not currently on immunosuppressive drugs such as chemotherapy, oral or parenteral prednisone or Tumor Necrosis Factor-alpha (TNF-α) inhibitor therapy.
* Not allergic to chicken/egg protein.
* Willing to have blood drawn (4 times) during the study.
* Willing to complete a simple diary documenting toxicity, pill count and any side effects of the medication and any reported illnesses during this period.
* Willingness to take 4 capsules per day, keep a symptom and capsule diary, and return these materials to the clinic at the conclusion of the study.
* Willingness to avoid all over the counter nutritional supplements, probiotics, and yogurts containing probiotics during the duration of the study.
* Patients who have provided their written informed consent prior to participation in the study and have signed and dated an appropriate Health Insurance Portability and Accountability Act (HIPAA) authorization form.
* Blood laboratory results within the 7 days of starting study drug
* Normal liver function as shown by:
* serum AST within upper limits of normal
* Adequate renal function as shown by :
* serum creatinine ≤ 2.0 mg/dL
* Hemoglobin > 11gm/dL; WBC: > 3.5X109 /L and platelets > 100 X 109 /L

Exclusion Criteria:

* Antibiotic use - current or within 2 weeks prior to start of the study.
* Chicken/Egg hypersensitivity or hypersensitivity to influenza vaccine components such as bactopeptone, beta-propiolactone, neomycin, gentamicin, monosodium glutamate, formaldehyde or formalin, gelatin, polyethylene glycol p-iso-octylphenyl ether (Triton X-100), polymyxin B, polyoxyethylene 9-10 nonyl phenol (Triton N-101, octoxynol 9), or thimerosal.
* Talc allergy
* Influenza vaccine within the prior 12 months.
* Immunosuppressed status either from illness such as acquired immunodeficiency syndrome (AIDS), or with concomitant chemotherapy, or iatrogenic immunosuppression such as prednisone or other drugs such as TNF-α inhibitor therapy.
* History of known serious illness such as active cancer (except localized skin or non-metastatic prostate cancer), poorly controlled congestive heart failure, poorly controlled diabetes, acute or progressive renal or hepatic failure, chronic obstructive lung disease requiring oxygen.
* Ongoing anti-influenza therapy with amantadine, rimantadine, oseltamivir or zanamivir
* Active or recent (within last 6 months) history consistent with acute influenza illness. Febrile illness with headache, sore throat and temperature more than 37.5C on the day of enrollment.
* Known chronic inflammatory bowel disease such as Crohn's disease, active bowel cancer (defined as being on chemotherapy or having an untreated bowel cancer)
* Hypersensitivity to any components of the AKSB, placebo or the vaccine.
* Oral typhoid vaccine use in the last 2 weeks.
* Patients who have participated in a clinical study and/or received any investigational medication during the last month (30 days) preceding study Day 1; or currently enrolled in an investigational study.
* Patients who, in the opinion of the investigator, possess insufficient mental or reading ability that prevents their understanding and providing informed consent and appropriate HIPAA authorization;
* Patients who, in the opinion of the Investigator, would not be able or willing to comply with the protocol;
* Patients who are unwilling or unable to comply with the study protocol for any other reason.
* History of Guillain-Barré Syndrome within 6 weeks following a previous dose of the inactivated vaccine.
* Allergy or contraindication to two or more of the following: vancomycin, penicillins, daptomycin, linezolid
* Allergy or contraindication to two or more of the following: fluconazole, deoxycholate amphotericin B, liposomal amphotericin B, itraconazole or voriconazole
* Blood laboratory results within the 7 days of starting study drug
* Abnormal normal liver function as shown by:
* serum AST above the upper limits of normal
* Impaired renal function as shown by :
* i. serum creatinine > 2.1 mg/dL
* Hemoglobin < 11gm/dL; WBC: < 3.5X109 /L and platelets < 100 X 109 /L

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
number of patients with adverse events | 127 days
  To evaluate the safety and tolerability of AKSB when administered with the influenza vaccine as compared to the influenza vaccine alone with placebo in patients ≥65 years of age.

SECONDARY OUTCOMES:
Compare stool presence of probiotic enterococcal strain | baseline to 21 days
  To evaluate for stool VRE presence pre-post intervention and to compare molecular fingerprinting of VRE isolated with the SF68 strain of enterococci used in the study drug to demonstrate safety of the study drug.
Immune response to Influenza A vaccine in the AKSB arm compare to Placebo | days 14, 28 days and 120 days after vaccination
  To determine whether AKSB can increase the protection rate [PR, (number of participants that achieve the protective antibody titer)] by 20% in the AKSB arm at days 14, 28 days and 120 days after vaccination among the elderly patients (≥ 65 years of age). Effect of age (65-75 years and >75 years), gender, underlying medical history and previous vaccination status (within the last 2 years) will evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Abinash Virk, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States